CLINICAL TRIAL: NCT06321965
Title: Characterization of New Phenotypes of Patients With Spinal Muscular Atrophy Treated With SMN Restoring Therapy
Acronym: PHENO SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0599
Record Dates: First submitted 2024-02-06; First posted 2024-03-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy
Keywords: Natural history; Spinal Muscular atrophy (SMA); Risdiplam; Onasemnogene abeparvovec; Nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Muscle Fatigue; Metabolism; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, multicenter, international study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMA patient treated with SRT (Experimental): Patients aged 0-15 with SMA type 1, 2 or 3, treated with TRS (nusinersen/risdiplam/onasemnogene abeparvovec/other).
  Interventions: Other: evaluation of muscle function; Other: First-line cognitive assessment; Other: second-line cognitive assessment; Other: Cardiac evaluation; Radiation: MRI; Other: Assessment of activity and muscle fatigue; Other: Assessment of bulbar function; Other: Evaluation of body composition and metabolism; Other: Questionnaires; Biological: Biocollection; Other: Skinfold measurement

INTERVENTIONS:
Other: evaluation of muscle function — Myogrip (≥ 6 years): precise dynamometric measurement of gripping force, measuring force in Newton up to 90kg with 0.01kg resolution. It's evaluated at D0, M6, M12, M18, and M24 Myopinch (≥ 6 years) : measure thumb-index force up to 15 kg with a resolution of 0.001 kg using a precision sensor equipped with two steel distance blades. It's evaluated at D0, M6, M12, M18, and M24
Other: First-line cognitive assessment — Vineland-II (All patients) : is a scale for assessing adaptive behaviors. will be carried out during the telephone call at M1/V2.
  All tests are evaluated at D0, and M18 :
  Bayley-4 language part (< 42 months) PVSE (≥ 4 years) CELF-5 (≥ 5 years) Conners-3 (≥ 6 years) AQ (≥ 4 years), EQ (≥ 11 years)
  M-CHAT-R (< 4 years) :
  SRS-2 (≥ 2 years)
Other: second-line cognitive assessment — In the event of positive cognitive screening at D0 or M18, a second-line cognitive assessment will be carried out at a subsequent visit. A list of tests is proposed below, but will be adapted according to the tests available at each center.
  * EVALO BB (0-2 years) or EVALO (2-6 years) or full CELF-5 (5-18 years) following positive screening in the communication domain of first-line tests (Vineland II communication domain, Bayley 4, CELF-5 pragmatic profile)
  * FEE and DSM-5 diagnostic criteria for ADHD (from age 6 only) following positive screening in the attention and executive functions domain of first-line tests (Conners 3, BRIEF)
  * M-CHAT-R/F (< 4 years) or SCQ (≥ 4 years) and ADOS-2 (≥ 12 years) following a positive screening in the area of social cognition and autistic traits on first-line tests (Vineland II, M-CHAT-R, SRS-2, EQ, AQ).
Other: Cardiac evaluation — All tests are evaluated at D0, M12, and M24 :
  Electrocardiogram (ECG) : This examination will be carried out in accordance with the 12 leads recording the following parameters: verification of sinus rhythm, P wave, PR interval, QRS complex (interval), ST segment, T wave, QT complex, heart rate.
  Cardiac ultrasound: Non-invasive ultrasound will focus on the following parameters measured from 2-dimensional images, to look for cardiomyopathy and/or structural abnormality:
  * end-diastolic/end-systolic diameter/left ventricular ejection fraction
  * Septal wall thickness / left ventricular posterior wall
  * Fractional shortening 24-hour Holter-ECG : This examination consists of a continuous test recording the heart rhythm for 24 hours.
Radiation: MRI — Cerebral MRI : Performed at D0, only for patients with ASI type 1 ≥ 6 years, or younger patients for whom the investigator considers that the examination can be performed without sedation or general anesthesia. It will include sequences:
  * 3D T1, gradient echo, 1.1 mm voxel, sagittal acquisition
  * axial T2, spin-echo, slice thickness 4 mm
  * 3D FLAIR, spin-echo, 1 mm voxel, sagittal acquisition Muscular MRI: performed at V1/J0, and V6/M24. The examination will include water-fat imaging (Dixon) in full-body, 3D mode, with proton density weighting and millimeter resolution.
Other: Assessment of activity and muscle fatigue — Syde® : evaluated at D0, M6, M12, M24. Patients aged 2 and over will receive the Syde® wearable device to collect their daily activities.
  Muscular endurance tests (≥ 6 years) : evaluated at D0, M12, M24 ( only one of 3 tests based on motor function level) oESNHPT : In this test, patients are asked to walk a 10-meter path. oESBBT : In this test, patients have to move 10 blocks over a partition. oESWT: In this test, patients must repeatedly place and remove 9 sticks in 9 holes.
  PedsQL Fatigue (≥ 2 years): evaluated at D0, M12, M24. Scale designed to measure fatigue in patients with acute and chronic conditions, as well as in healthy school and community populations.
  Fatigue rating scale (≥ 6 years): evaluated at D0, M12, M24. The fatigue assessment scale has 11 numerical points ranging from 0 to 10. The patient is asked to give a rating that best reflects his or her perception of fatigue at that particular moment.
Other: Assessment of bulbar function — DDD-pNMD (≥ 2 years) : evaluated at D0, M6, M12, M18, and M24, is a list of 9 questions used by doctors to screen for dysphagia and dysarthria.
  NdSSS (All Patients) : evaluated at D0, M6, M12, M18, and M24, is an 8-level scale for assessing swallowing.
  TOMASS-c : (≥ 4 years of age, in patients able to eat solids safely, after assessment of the risk of a false route by the speech therapist): this is a score designed to assess mastication when eating a cracker. Age-dependent standards exist for different types of cracker.
  - Fluid intake test (> 110 cm, in patients able to drink a liquid safely, after assessment of the risk of a false route by the speech therapist): swallowing limit.
Other: Evaluation of body composition and metabolism — Food survey : The dietary survey questionnaire will be sent to parents at D0 and M18. Parents will be asked to complete it for 3 days before the M6 and M24.
  Bioelectrical impedancemetry: Evaluated at M6 and M24. Renal ultrasound: Evaluated at M6, is a non-invasive examination that analyzes the appearance of the kidney and urinary tract.
  Dual-energy X-ray absorptiometry (DXA) : Evaluated at M6, it measures body composition using spectral imaging, including fat mass, lean mass and bone mineral density.
  Fibroscan : Evaluated at M6 and M24. This examination uses pulse elastography to measure liver elasticity, which provides information on the presence of hepatic fibrosis, and sound attenuation, which provides information on the presence of liver fat overload.
  Indirect calorimetry : Evaluated at M6. This device enables precise measurement of Resting Energy Expenditure , Respiratory Quotient and metabolic substrate oxidation.
Other: Questionnaires — SMAIS : The questionnaire has been developed specifically for ASI. At D0, M6, M12, M18 and M24.
  HUI2 : specializes in preference-based measures of health-related quality of life. At D0, M6, M12, M18 and M24.
  Peds QL : is a modular instrument designed to measure health-related quality of life and disease-specific symptoms. At D0, M6, M12, M18 and M24.
  Neuromuscular module : 17 disease-related items. It is evaluated at D0, M6, M12, M18 and M24.
  Family impact module : It measures parents' reported physical, emotional, social and cognitive functioning, communication and concerns. At D0, M12, and M24.
  ASI cost questionnaire: At visit 1 (D0): This questionnaire, completed by the parents, includes information on occupation, parents' working hours and any reduction in them due to the child's pathology, the number of working days missed by the parents or school days missed by the child, and disability-related costs.
Biological: Biocollection — A blood bio collection (optional) will be offered to patients at D0, M6 , M12, M18, M24.
  Patients receiving intrathecal injections will also be offered the opportunity to participate in a CSF (cerebrospinal fluid) biocollection (optional).
Other: Skinfold measurement — The tricipital point should be marked on the posterior aspect of the arm, on the midline of the tricipital muscle, midway between the acromion and the radius. At D0, M6, M12, M18 and M24

SUMMARY:
With the advent of new treatments for ASI, new phenotypes are emerging. The investigators propose to describe these new phenotypes by prospectively following children with ASI of all types treated with TRS and aged under 16 for 2 years.

The investigators also propose to evaluate potential assessment tools to determine whether they are relevant for monitoring this population, either routinely or for future clinical trials. The investigators also aim to collect the total costs associated with ASI in order to propose a first prospective medico-economic study in France.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed infantile or juvenile spinal muscular atrophy
* Treated with a therapy that restores SMN protein expression (e.g. nusinersen, risdiplam, onasemnogene abeparvovec)
* Aged 0 to 15 years inclusive
* Informed consent signed by both parent(s)/legal guardian(s) and patient's assent
* Affiliated or beneficiary of a health insurance plan*. * for inclusion in France

Exclusion Criteria:

* Other condition likely to interfere significantly with ASI assessment and clearly unrelated to the disease
* Other associated neurological disease
* Current pregnancy or breast-feeding (a pregnancy test will also be performed at inclusion).

Please note that patients with a specific contraindication to MRI (i.e. metallic foreign body, claustrophobia and other reasons determined by the investigators) will be allowed to participate in the study, but MRI will not be performed.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2029-01-24 (Estimated); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Markers of disease progression and description of different phenotypes, at : muscular and functional | Every 6 months from inclusion (Day 0, Month6, Month12, Month18, Month24)
  A composite score indicating the overall motor development trajectory for patients from study inclusion to Month 24 (M24).
  Calculation: Assign numerical values or categories to represent the motor development stages, with higher scores indicating positive development and lower scores indicating decline.
Markers of disease progression and description of different phenotypes, at : muscular and functional | Every 6 months from inclusion (Day 0, Month 6, Month 12, Month 18, Month 24)
  The trajectory of mean scores for motor function and muscle strength measured using CHOP-INTEND for patients aged 0-2 years. Scores are assessed every 6 months from inclusion (Day 0, Month 6, Month 12, Month 18, Month 24).
  Scale: CHOP-INTEND scale (0-64) Minimum Value: 0 Maximum Value: 64 Interpretation: Higher scores indicate improved motor function and muscle strength.
Markers of disease progression and description of different phenotypes, at : muscular and functional | Every 6 months from inclusion (Day 0, Month 6, Month 12, Month 18, Month 24)
  Motor Function Measure 32 (MFM-32), is a quantitative scale created to measure global motor functional abilities in a person with neuromuscular disease. It contains 32 items, each marked from 0 to 3. The total score and the sub-scores are expressed as a percentage of the maximum possible score.
  Scale Range: 0 to 100 (Minimum to Maximum Values)
  Interpretation: Higher scores on the Motor Function Measure 32 (MFM-32) indicate improved motor function and muscle strength.
  The lower the total score, the more severe the impairment.
Markers of disease progression and description of different phenotypes, at : muscular and functional | Every 6 months from inclusion (Day 0, Month 6, Month 12, Month 18, Month 24)
  Motor function and muscle strength: Trajectory of mean score between inclusion and M24: 6-minute walk test (≥ 6 years walking)
Markers of disease progression and description of different phenotypes, at : muscular and functional | Every 6 months from inclusion (Day 0, Month 6, Month 12, Month 18, Month 24)
  Motor function and muscle strength: Trajectory of mean score between inclusion and M24:
  Myogrip (≥ 6 years), Myopinch (≥ 6 years)
Markers of disease progression and description of different phenotypes, at : Fatigue | Syde: At Day 0, Month 6, Month 12 and Month 24
  For All:
  Upper limb kinematics and power
  For Walkers:
  Gait variables, arm swing variables, walking perimeter Interpretation: Specific statistical quantities related to upper limb kinematics and power, and additional variables for walkers.
  Calculation: Analyze statistical quantities at each time point for Syde
Markers of disease progression and description of different phenotypes, at : Fatigue | Endurance test (≥ 6 years)
  Endurance time from 0 to 1200 The primary outcome measure for fatigue-related markers involves the endurance test (≥ 6 years), specifically assessing ESNHPT, ESBBT, and ESWT. The primary focus is on the proportion of patients who stop before completing the test (yes/no) and, if applicable, the mean time to stop in seconds.
  ESNHPT: Endurance Test - Non-Handheld Propulsion Task ESBBT: Endurance Test - Bodyweight Bearing Task ESWT: Endurance Test - Walking Task
Markers of disease progression and description of different phenotypes, at : Fatigue | at Day 0, Month 12 and Month 24
  Pediatric Quality of Life Inventory (PedsQL) Fatigue Total Score Minimum Value: 0 Maximum Value: 24 Interpretation: A higher score within the range indicates increased fatigue, while a lower score suggests less fatigue.
Markers of disease progression and description of different phenotypes, at Orthopaedic level | Joint amplitudes at Day 0, Month 6, Month 12 and Month 24
  Joint amplitudes: Trajectory of joint amplitude changes (angle) between Day 0 and Month 24 for each location:
  Hip (right and left), Knee (right and left), Ankles, Elbow, Wrist, Long fingers.
Markers of disease progression and description of different phenotypes, at Orthopaedic level | Clinic and spinal radiography at Day 0, Month 12,Month 18, Month 24
  (For Non-Operated Patients): Presence or Absence of Radiological Scoliosis
Markers of disease progression and description of different phenotypes, at Orthopaedic level | at Day 0, Month 24+/- Month 6, Month 12, Month 18
  Clinical and pelvic radiography:
  Proportion of patients with hip eccentricity (>10% on Reimers index) at Day 0 and Month 24
Markers of disease progression and description of different phenotypes, at the cognitive level: Vineland-II | At Month 1
  Vineland II Adaptive Behaviour scales (VABS) total mean score and subscale mean scores.
  Standardized questionnaire filled by the Neupsy during an interview with the parents or the patient himself if possible. 5 domains. Maximum score 160, minimum score 20, mean score 100, standard deviation 15
Markers of disease progression and description of different phenotypes, at the cognitive level: Bayley-4 | At Day 0 and Month 18
  Bayley-4 Scales of Infant and Toddler Development is standardized developmental assessment tool for determining a child's developmental status at a given age (up to 42 months) BAYLEY-4 assess development in children of 1-42 months old in 5 domains: cognition, motor, language, socio-emotional, and adaptive behavior.
  The Bayley-4 raw scores from 0-84 for the receptive communication subtest, 0-74 for the expressive communication subtest a higher score denotes a better outcome. The Bayley-4 standard score norms are converted to percentiles from <0.1 to >99.9 for the language
Markers of disease progression and description of different phenotypes, at the cognitive level: BRIEF (Behavioral Rating Inventory of Executive Function) | At Day 0 and Month 18
  BRIEF provides scores that are used to evaluate different aspects of executive function. The scores are typically presented in various subscales, each focusing on a specific domain of executive function.
  composite T-score for overall developmental function equal to or greater than 65 (-1.5 SD)
  The " composite T-score for overall developmental function equal to or greater than 65 (-1.5 SD)" indicates that a T-score composite for the overall developmental function is considered elevated or clinically significant if it equals or exceeds 65, which is 1.5 standard deviations above the mean in a standardized population. Higher scores on the BRIEF suggest greater difficulties in executive functioning, with a T-score of 65 or above indicating a higher level of impairment or challenges in this domain.
Markers of disease progression and description of different phenotypes, at the cognitive level: Conners-3 | At Day 0 and Month 18
  - CONNERS-3 : 108-item hetero-questionnaire to assess the presence of symptoms of inattention, hyperactivity, impulsivity and other frequently associated disorders in children and adolescents aged 6 to 18. Symptoms are rated on a Likert scale with severity ratings from 0 (not at all/never) to 3 (very much/ very frequently). The Conners t-score range from 0 - 100. The higher the number, the worse the outcome
Markers of disease progression and description of different phenotypes, at the cognitive level: CELF-5 (Language and communication assessment battery) | At Day 0 and Month 18
  Standard Score: This score are derived from the total raw scores for each test and are on a normalized score scale that has a mean of 10 and a standard deviation (SD) of 3
  The mean score is 100, with a standard deviation of 15, meaning:
  that standard scores between 85-115 are within the normal range. Score Mild: 70-85, Moderate: 55-70, Severe: 55 and lower
Markers of disease progression and description of different phenotypes, at the cognitive level: EQ (Empathy quotient), AQ (Autism Quotient) | At Day 0 and Month 18
  Evaluation of the French Version of Screening Questionnaires for Autism and Asperger Syndrome: Autism Spectrum Quotient (AQ) Empathy Quotient (EQ) EQ is a 40-item questionnaire designed to measure empathy for patients aged 11 and above. The maximum score for this questionnaire is 80.
  Threshold score: ↓30 . Scores of 30 or less indicate a lack of empathy common in people with Autism.
  AQ comprises 50 questions, with 5 groups of 10 questions assessing imagination, social skills, attention switching, attention to detail and communication skills. Each of these items scores 1 point if the respondent records abnormal or autistic like behaviour. The minimum score on the AQ is 0 and the maximum 50 with high scores indicating high autistic traits.
Markers of disease progression and description of different phenotypes, at the cognitive level: M-CHAT-R (Modified Checklist for Autism in Toddlers) | At Day 0 and Month 18
  The Modified Checklist for Autism in Toddlers, Revised (M-CHAT-R) is a screener that will ask a series of 20 questions about the child's behavior.
  To score the M-CHAT-R, we add up the number of at-risk responses, and follow the algorithm below:
  LOW RISK:
  Total score between 0 and 2
  MEDIUM RISK:
  Total score between 3 and 7
  HIGH RISK:
  Total score between 8 and 20
Markers of disease progression and description of different phenotypes, at the cognitive level: SRS-2 (Social Responsiveness Scale, Second Edition) | At Day 0 and Month 18
  SRS measures social ability of children from 2 years to 18 years old. It is used primarily with individuals with Autism Spectrum Disorder (ASD), family members of individuals with ASD, and others who have social impairments. Parent or teacher questionnaire (65 items on a 4-point Likert scale). High scores are associated with more severe social impairments.
  Raw total scores are converted to gender-normed T scores
  SRS-2 total T-scoring:
  * Less than or equal to 59 = Within normal limits (generally not associated with ASD)
  * Between 60-65 = Mild range
  * Between 66-75 = Moderate range
  * Greater than or equal to 76 = Severe range (strongly associated with clinical diagnosis of ASD)
Markers of disease progression and description of different phenotypes, at the cognitive level: PVSE (Basic visuo-spatial perception) | At Day 0 and Month 18
  - Proportion of patients with overall score:
  * < OL_inf
  * OL_inf ≤ x < Q1
  * Q1 ≤ x < M
  * M ≤ x < Q3
  * Q3 ≤ x < Q3
  * ≥ OL sup
Markers of disease progression and description of different phenotypes, at the brain level | At Day 0
  Cerebral MRI :
  Proportion of patients with :
  * Posterior fossa anomaly
  * Midline anomaly
  * White matter anomaly
  * Cortical anomaly
  * Basal ganglia anomaly
  * Ventricular system anomaly
  * Pericerebral space abnormality
  * Brain MRI abnormality (including above variables)
Markers of disease progression and description of different phenotypes, at Cardiology level | At Day 0 +/- Month 12, Month 24
  Electrocardiogram (ECG): An abnormal ECG, with proportion for each type of abnormality Holter-ECG: An abnormal Holter-ECG, with proportion for each type of abnormality Echocardiography (only if troponin anomaly): Abnormal echocardiography, with proportions for each type of abnormality
Markers of disease progression and description of different phenotypes, at metabolic level : Anthropometric measurement trends | Anthropometric measurements at Day 0, Month 6, Month 12, Month 18, Month 24
  Anthropometric measurements may be used to monitor growth and nutritional status.
  Outcome of tracking these measurements could be the identification of trends related to weight gain and muscle mass development. Assessing changes in weight and body composition over time can provide valuable insights into the impact of SMA on physical development, guide nutritional interventions, and help healthcare providers tailor supportive care to address the unique needs of children with SMA
Markers of disease progression and description of different phenotypes, at metabolic level : | Food survey at Month 6, Month 24
  Food survey: average food intake
Markers of disease progression and description of different phenotypes, at metabolic level : fractures | at Day 0, Month 6, Month 12, Month 18, Month 24
  Number of fractures by location and mechanism
Markers of disease progression and description of different phenotypes, at metabolic level : renal ultrasound | at Month 6
  Proportion of patients with abnormal renal ultrasound
Markers of disease progression and description of different phenotypes, at metabolic level : Absorptiometry (DXA) | at Month 6
  DXA measurement will be performed to assess patient's body composition.
  Average values + SD (Standard Deviation):
  Lean mass and fat mass (kg) with deficit or excess of lean mass and fat mass (%) Total bone mineral content (g) Bone mineral density (z-score) at the spine, femoral neck, and distal femur
Markers of disease progression and description of different phenotypes, at metabolic level: Calorimetry | at Month 6
  Potential outcome of using this device is the accurate measurement of Resting Energy Expenditure (REE). This information can be particularly important in managing the nutritional needs of individuals with SMA, helping healthcare providers optimize dietary plans to meet the specific energy requirements of patients dealing with this neuromuscular disorder. Resting Energy Expenditure (REE).
Markers of disease progression and description of different phenotypes, at metabolic level : Impedancemetry | at Month 6 and Month 24
  Average +SD values of Impedancemetry results
Markers of disease progression and description of different phenotypes, at metabolic level : Fibroscan | At Month 6 and Month 24
  The FibroScan result is reported in kilopascals (kPa), representing the liver stiffness. The numerical value indicates the degree of stiffness, which correlates with the extent of liver fibrosis. The interpretation of the FibroScan score is as follows:
  Low Stiffness (Low kPa): Indicates a healthier, less fibrotic liver.
  Intermediate Stiffness: May suggest some degree of fibrosis, and further evaluation may be needed to determine the extent.
  High Stiffness (High kPa): Indicates more advanced liver fibrosis or cirrhosis.
Markers of disease progression and description of different phenotypes, at biological analysis | At Day 0, Month 6, Month 12, Month 18, Month 24
  Proportion of patients with biological abnormalities for each parameter:
  Blood/platelet count: Hb, leukocytes, platelets, ASAT, ALAT, GGT, PAL, TP, Sodium, potassium, bicarbonates, calcium, phosphorus, creatinine, glucose, proteins, urea, cystatin C, Troponin, BNP, NT-pro-BNP, Iron, Ferritin, copper, zinc, selenium, magnesium, Vitamins A,C,D,E, B12, Folates, Albumin, prealbumin, retinol-binding protein, ultra-sensitive C-reactive protein (CRP), FibroTest, PTH (parathormone) For these patients : % above normal
  * above
  * or below
Markers of disease progression and description of different phenotypes, at In terms of quality of life and autonomy | PedsQL family impact at Day 0, Month 12, Month 24
  Score evolution trajectory :
  PedsQL (Pediatric Quality of Life Inventory™) family impact The 36-item PedsQL™ Family Impact Module Scales encompass 6 scales measuring parent self-reported functioning: 1) Physical Functioning (6 items), 2) Emotional Functioning (5 items), 3) Social Functioning (4 items), 4) Cognitive Functioning (5 items), 5) Communication (3 items), 6) Worry (5 items), and 2 scales measuring parent-reported family functioning; 7) Daily Activities (3 items) and 8) Family Relationships (5 items).
  Scale Scores are computed as the sum of the items divided by the number of items answered.
  higher scores indicate better functioning (less negative impact)
Markers of disease progression and description of different phenotypes, at In terms of quality of life and autonomy | HUI-2, generic PedsQL and neuromuscular module at Day 0, Month 6, Month 12, Month 18 and Month 24
  HUI2 classification system consists of attributes (domains) of health to 6 levels of functional ability/disability within each attribute. For each attribute, singleattribute utility functions range from 0.00 for highly disabled (deaf) to 1.00 Score total : 0 - 1
Markers of disease progression and description of different phenotypes, at respiratory level : Chest/head circumference ratio (PT/PC ratio) (up to 3 years) | at Day 0, Month 6, Month 12, Month 18 and Month 24
  Outcome measure related to hospitalizations in the context is "Proportion of Patients with Escalation of Respiratory Assistance." This measure assesses the percentage of patients who experienced an escalation in respiratory support during their hospital stay, encompassing variables such as increased settings on home machines, use of resuscitative NIV, or intubation. This outcome provides critical insights into the respiratory management and support needs of patients during their hospitalizations.
Markers of disease progression and description of different phenotypes, at respiratory level : Chest/head circumference ratio (PT/PC ratio) | at Day 0, Month 6, Month 12, Month 18 and Month 24
  Evolution of the PT/PC ratio trajectory
Markers of disease progression and description of different phenotypes, at respiratory level : O2 saturation and nocturnal TcPCO2 | at Day 0, Month 12, Month 24
  Evolution trajectory: This measure focuses on the percentage of children experiencing elevated levels of transcutaneous carbon dioxide (TcPCO2), specifically defined as time spent with TcPCO2 levels exceeding 50mmHg. This outcome is crucial in assessing the severity of respiratory compromise and may guide interventions to address and manage hypercapnia in the pediatric population.
Markers of disease progression and description of different phenotypes, at respiratory level: Respiratory function tests (≥ 6 years) | at Day 0, Month 12, Month 24
  Evolutionary trajectory: Evolution of Inspiratory Vital Capacity in Different Positions (% of Theoretical). This measure assesses changes over time in the percentage of theoretical inspiratory vital capacity achieved while standing or sitting and while lying down. This outcome provides valuable information about respiratory muscle function and potential changes in the ability to generate inspiratory volumes in different body positions.
Markers of disease progression at respiratory level | points (Day 0, between Day 0-Month 12, between Month 12 and Month 24)
  Evolutionary trajectory :
  Proportion of patients with central sleep apnea syndrome Proportion of patients with obstructive sleep apnea syndrome Proportion of patients with alveolar hypoventilation syndrome
Markers of disease progression and description of different phenotypes, at bulbar level (Evaluation of dysphagia and dysarthria): DDD-pNMD (Diagnostic list for Dysphagia and Dysarthria in pediatric NeuroMuscular Disorders) | At Day 0, Month 6, Month 12, Month 18, Month 24
  The DDD-pNMD is a scale where items are scored by a Speech-Language Therapist (SLT) on a 4-point scale, ranging from 0 (normal) to 3 (severe problems/impossible). The scale is designed to assess various aspects of swallowing and speech in children with neurological conditions.
  The DDD-pNMD screening is positive if score greater than or equal to 1.
Markers of disease progression and description of different phenotypes, at bulbar level (Evaluation of dysphagia and dysarthria): NdSSS (Neuromuscular Disease Swallowing Status Scale). | At Day 0, Month 6, Month 12, Month 18, Month 24
  An 8-stage Neuromuscular Disease Swallowing Status Scale (NdSSS) Positive if the level on the NdSSS scale is less than or equal to 7
Markers of disease progression and description of different phenotypes, at the level of Characteristics at inclusion: age of patient | At Day 0
  + SD: Age, age of onset of symptoms, age at start of treatment
Markers of disease progression and description of different phenotypes, at the level of Characteristics at inclusion : patient gender | At Day 0
  Proportion of male patients
Markers of disease progression and description of different phenotypes, at the level of Characteristics at inclusion: SMA TYPE | At Day 0
  Proportion of patients by type of SMA (1, 2, 3) and by treatment
Markers of disease progression and description of different phenotypes, at the level of Characteristics at inclusion: number of copy | At Day 0
  SMN2 copy number distribution
Markers of disease progression and description of different phenotypes, at the level of Characteristics at inclusion: treatment | At Day 0
  Calculate the proportion of patients who underwent treatment changes, expressed as a percentage of the total study population.This measure provides insights into the adaptability and potential issues with the current therapeutic approach or side effects.
  A higher proportion of treatment changes may prompt further investigation and adjustments in treatment protocols, aiming to enhance overall patient outcomes.
  This focused outcome measure aims to capture the essence of treatment dynamics within the SMA patient population.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Pediatric Rehabilitation Service - L'Escale Mother and Child Hospital, Bron, Rhone
  - CHRU of Brest, Brest
  - Pediatric Neurology and Resuscitation Raymond-Poincare Hospital, Garche
  - Pediatric Neurology Swynghedauw Hospital, Lille
  - Marseille University Hospital - Timone Hospital Department of Pediatric Neurology - Specialized Pediatrics and Child Medicine, Marseille
  - I-Motion Pediatric Clinical Trial Platform Armand Trousseau Hospital, Paris
  - Hautepierre Hospital - Mother and Child Hospital, Strasbourg
  - Department of Pediatrics - Neurology and Infectious Diseases Toulouse University Hospital - Children's Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No